CLINICAL TRIAL: NCT04584216
Title: Evaluation of the Effects and Safety by the Steam Eye Mask With Acupoints Stimulation for VDT User
Brief Title: Effects and Safety of Steam Eye Mask With Acupoints Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kao (Taiwan) Corporation (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Kao-001
Record Dates: First submitted 2020-09-28; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Dry Eye Symptom; Eye Fatigue
Keywords: Steam Eye Mask; Acupoints Stimulation; Dry Eye Symptom; Eye Fatigue; Visual Display Terminal; Moist Heat; Massage
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steam Eye Mask With Acupoints Stimulation (Experimental): The Steam Eye Mask with acupoints stimulation (SEM with acupoints stimulation), is an eye mask which contains iron (Fe) and generates the heat with the steam (the moist heat) by the oxidative reaction of the iron with oxygen in air.
  Also, on the eyebrow have the acupoints made by nonwoven fabric can use hands to massage.
  The temperature of the moist heat is approximately 40 degree C and the moist heat lasts for around 20 minutes and use hands to massage the acupoints on the eyebrows for the first 3 minutes.
  Interventions: Other: Steam Eye Mask with acupoints stimulation
- Steam Eye Mask (Active Comparator): The Steam Eye Mask (SEM), is an eye mask which contains iron (Fe) and generates the heat with the steam (the moist heat) by the oxidative reaction of the iron with oxygen in air.
  The temperature of the moist heat is approximately 40 degree C and the moist heat lasts for around 20 minutes.
  Interventions: Other: Steam Eye Mask

INTERVENTIONS:
Other: Steam Eye Mask with acupoints stimulation — A participant needs to use SEM with acupoints stimulation once a day for 10 days and use hands to massage the acupoints on the eyebrows for the first 3 minutes, total application time at least for 20 minutes.
  Other Names: SEM with acupoints stimulation
  Arms: Steam Eye Mask With Acupoints Stimulation
Other: Steam Eye Mask — A participant needs to use SEM once a day for 10 days, total application time at least for 20 minutes.
  Other Names: SEM
  Arms: Steam Eye Mask

SUMMARY:
To evaluate the effects and safety of the steam eye mask with acupoints stimulation by the moist heat of approximately 40 degree C for 20 minutes and massage acupoints on eyebrows for eye fatigue, dry eye symptoms and symptom-induced decline of Quality of life (QoL) in VDT users.

DETAILED DESCRIPTION:
A prospective study is conducted to evaluate the effect of the steam eye mask with acupoints stimulation on eye fatigue and dry eye symptoms in VDT users. The effects and safety of the single therapy by the moist heat of approximately 40 degree C for 20 minutes with eyebrows acupoints massage for the first 3 minutes are evaluated in the single application study, and the effects and safety of the repeated therapy by the moist heat applied and massage acupoints on eyebrows once per working day for two weeks are evaluated in the repeated application study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged from 20 to 69 years old (both inclusive).
2. Participants who use VDTs, including laptops, electronic tablets, readers and smartphones for 6 hours or more a day.
3. Participants who respond to the 16 symptoms of visual symptoms related to computer use in the working population for the total score over 6 based on a computer vision syndrome questionnaire.
4. Participants who respond to more than 1 of 12 typical dry eye symptoms by "constantly" or "often" based on a dry eye questionnaire.
5. Participants are able and willing to comply with all protocol requirements and procedures.
6. Participants who must be capable of providing informed consent document, with one's signature.

Exclusion Criteria:

1. Participants with eye diseases that could affect the ocular surface (e.g. Ocular inflammation, infectious conjunctivitis, allergic diseases, autoimmune diseases and collagen diseases).
2. Participants who have been treated by physicians because of eye diseases and do not recover from that disease yet at the moment of joining to this study, or participants who need to be treated by physicians because of eye disease.
3. Participants with the excessive meibomian lipid secretion (seborrheic MGD).
4. Participants with trauma, swelling and eczema at the skin around eyes.
5. Participants with allergic reaction for heating, abnormality of the heat or depression of the heat.
6. Participants who are deemed inappropriate to participate in this study by physicians.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Assessment of symptoms and mood state (Visual Analog Scale, VAS) evaluated by participants. | 14 days
  The severity of symptoms and mood state are evaluated using a VAS by each participant. A VAS is a horizontal line, 100mm in length, anchored by word descriptors at each end. Participants mark on the line the point that they feel their perception of their current state. The VAS score is determined by measuring the length from the left hand end of the line to the point that they mark. The five symptoms to be evaluated are: tiredness of eyes, dryness of eyes, grittiness of eyes, blurred vision, and ocular discomfort. Each symptom is relieved as the VAS score decreases. The mood states to be evaluated are: relaxation and comfort. Each mood state is enhanced as the VAS score increases.

SECONDARY OUTCOMES:
The computer visual syndrome questionnaire (CVS-Q) evaluated by participants. | 19 days
  The computer vision syndrome questionnaire (CVS-Q) is applied to evaluate the visual health of workers exposed to the computer screen. This questionnaire consists of sixteen items with the response options of the severity (frequency and intensity) of each particular symptom and the overall symptom severity (CVS score). The score of each ocular discomfort is calculated by the frequency multiplies the intensity. The frequency for each symptom is answered by the subject as never, occasionally, and often/always which are coded as 0, 1, and 2, respectively. The intensity is defined for two options as 1 for moderate and 2 for intense, respectively. Moreover, the score obtained for each item will then be coded as 1 while the multiplied score is 1 or 2; and 2 while the multiplied score is 4. The results can be compared between different individuals or in the same individual at different times and circumstances. The higher score a subject gained, the worsen ocular condition he/she experienced.
Dry eye questionnaire evaluated by participants. | 19 days
  The dry eye questionnaire will be used for evaluate the dry eye symptom of each participant. This questionnaire consists of 12 typical dry-eye-related symptoms, include 1. Ocular fatigue, 2. Discharge, 3. Foreign body sensation, 4. Heavy sensation, 5. Dry sensation, 6. Uncomfortable sensation, 7. Excess tearing, 8. Blurred vision, 9. Itching, 10. Sensitivity to bright light, 11. Redness, 12. Pain. Each symptom will be evaluated from never, sometimes, often, and Constantly.
The quality of life (Dry-Eye-Related Quality of Life Score, DEQS) evaluated by participants. | 14 days
  The Dry-Eye-Related Quality of Life Score can assess various aspects of Quality of Life including its mental aspect. This questionnaire consists of 15 items related to dry eye symptoms(0 to 4, 0 as never, the less score as mild) and influence(1-4, the less score as rare) on daily life, and the overall degree of Quality of Life Score impairment is calculated as a summary score. The subject also grades the overall for the past week, including subject's eye symptoms and how they have affected subject's daily life, it will be graded from 1 to 6, the lower score means the subject is in better condition. DEQS score is decreased as Quality of Life Score is improved.
Measurement of Tear Meniscus Height (TMH) using Oculus Keratograph 5M by an examiner. | 14 days
  Tear Meniscus Height is observed with Oculus Keratograph 5M.
Tear film breakup time (TBUT) evaluated by an examiner. | 14 days
  Tear film breakup time is the parameter of tear film stability, defined as the time to initial breakup of the tear film after a blink.
Schirmer test evaluated by an examiner. | 19 days
  Schirmer test is an estimation of tear flow reflex by insertion of a filter paper into the conjunctival sac. This test is performed with the participants' eyes closed in 5 minutes.
Meibomian gland expression evaluated by an examiner. | 19 days
  Meibomian gland expression can be performed as an indicator of meibomian gland function, meibum expressibility and quality. The secretion expressed from the glands is observed with a physical force applied to the outer surface of the eyelid to determine whether a specific meibomian gland is functional and capable of providing secretion.
Visual acuity (VA) evaluated by an examiner. | 14 days
  The normal visual acuity is measured for both eyes separately using a Snellen chart.
Intraocular pressure (IOP) evaluated by an examiner. | 14 days
  The intraocular pressure is measured for both eyes separately using the tonometer.
Ocular surface/eyelids findings diagnosed by an examiner. | 19 days
  An ophthalmologist observes the cornea, conjunctiva, and eyelids for each participant and confirms whether there are any inflammation and hyperemia on the ocular surface or any other abnormalities on the ocular surface and eyelids before and after the application of IP.
  The slit lamp is applied to evaluate the following 6 items for both eyes including 1. Lid Margin Irregularity, 2. Lid Margin Vascularity, 3. Meibomian Orifice Plugging, 4. Mucocutaneous J Retroplacement, 5. Surface Finding Cornea, and 6. Surface Finding Conjunctiva. And the clinical judgments of normal or abnormal among these items will then assess by the investigators.
Diary reported by a participant. | 14 days
  Participants are asked to record the time, date, place and adverse events, if there is, in a daily questionnaire after every use of IP. If there is any report of adverse events, an ophthalmologist determines the severity and the relationship of the adverse events to using IP.
Adverse events | 19 days
  All adverse events will be record, and the incidence rates will be calculated.
Staining of ocular surface evaluated by an examiner | 14 days
  Ocular surface damage is assessed by staining cornea and conjunctiva. The liquid of fluorescein is instilled by the micropipette to stain the ocular surface. The staining of ocular surface is graded on a scale of 0 to 3 on the cornea and both areas of the conjunctiva, and then summed (Total range in 0-9 points) for each eye, according to the van Bijsterveld system.

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Shiou Hwang, M.D.,Ph.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kao (Taiwan) Corporation, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cushman WH. Reading from microfiche, a VDT, and the printed page: subjective fatigue and performance. Hum Factors. 1986 Feb;28(1):63-73. doi: 10.1177/001872088602800107. No abstract available. PMID 3710486
- [Background] Uchino M, Yokoi N, Uchino Y, Dogru M, Kawashima M, Komuro A, Sonomura Y, Kato H, Kinoshita S, Schaumberg DA, Tsubota K. Prevalence of dry eye disease and its risk factors in visual display terminal users: the Osaka study. Am J Ophthalmol. 2013 Oct;156(4):759-66. doi: 10.1016/j.ajo.2013.05.040. Epub 2013 Jul 24. PMID 23891330
- [Background] Lin PY, Tsai SY, Cheng CY, Liu JH, Chou P, Hsu WM. Prevalence of dry eye among an elderly Chinese population in Taiwan: the Shihpai Eye Study. Ophthalmology. 2003 Jun;110(6):1096-101. doi: 10.1016/S0161-6420(03)00262-8. PMID 12799232
- [Background] Skilling FC Jr, Weaver TA, Kato KP, Ford JG, Dussia EM. Effects of two eye drop products on computer users with subjective ocular discomfort. Optometry. 2005 Jan;76(1):47-54. doi: 10.1016/s1529-1839(05)70254-2. PMID 15682562
- [Background] Odaka A, Toshida H, Ohta T, Tabuchi N, Koike D, Suto C, Murakami A. Efficacy of retinol palmitate eye drops for dry eye in rabbits with lacrimal gland resection. Clin Ophthalmol. 2012;6:1585-93. doi: 10.2147/OPTH.S35584. Epub 2012 Oct 1. PMID 23055683
- [Background] Mori A, Shimazaki J, Shimmura S, Fujishima H, Oguchi Y, Tsubota K. Disposable eyelid-warming device for the treatment of meibomian gland dysfunction. Jpn J Ophthalmol. 2003 Nov-Dec;47(6):578-86. doi: 10.1016/s0021-5155(03)00142-4. PMID 14636848
- [Background] Abramson DI, Tuck S Jr, Lee SW, Richardson G, Levin M, Buso E. Comparison of wet and dry heat in raising temperature of tissues. Arch Phys Med Rehabil. 1967 Dec;48(12):654-61. No abstract available. PMID 6073416
- [Background] Geerling G, Tauber J, Baudouin C, Goto E, Matsumoto Y, O'Brien T, Rolando M, Tsubota K, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on management and treatment of meibomian gland dysfunction. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2050-64. doi: 10.1167/iovs.10-6997g. No abstract available. PMID 21450919
- [Background] Segui Mdel M, Cabrero-Garcia J, Crespo A, Verdu J, Ronda E. A reliable and valid questionnaire was developed to measure computer vision syndrome at the workplace. J Clin Epidemiol. 2015 Jun;68(6):662-73. doi: 10.1016/j.jclinepi.2015.01.015. Epub 2015 Jan 28. PMID 25744132
- [Background] Toda I, Fujishima H, Tsubota K. Ocular fatigue is the major symptom of dry eye. Acta Ophthalmol (Copenh). 1993 Jun;71(3):347-52. doi: 10.1111/j.1755-3768.1993.tb07146.x. PMID 8362634
- [Background] Sakane Y, Yamaguchi M, Yokoi N, Uchino M, Dogru M, Oishi T, Ohashi Y, Ohashi Y. Development and validation of the Dry Eye-Related Quality-of-Life Score questionnaire. JAMA Ophthalmol. 2013 Oct;131(10):1331-8. doi: 10.1001/jamaophthalmol.2013.4503. PMID 23949096
- [Background] The epidemiology of dry eye disease: report of the Epidemiology Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):93-107. doi: 10.1016/s1542-0124(12)70082-4. PMID 17508117
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Methodologies to diagnose and monitor dry eye disease: report of the Diagnostic Methodology Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):108-52. doi: 10.1016/s1542-0124(12)70083-6. PMID 17508118
- [Background] Shimazaki J, Sakata M, Tsubota K. Ocular surface changes and discomfort in patients with meibomian gland dysfunction. Arch Ophthalmol. 1995 Oct;113(10):1266-70. doi: 10.1001/archopht.1995.01100100054027. PMID 7575257
- [Background] Bron AJ, Benjamin L, Snibson GR. Meibomian gland disease. Classification and grading of lid changes. Eye (Lond). 1991;5 ( Pt 4):395-411. doi: 10.1038/eye.1991.65. PMID 1743355
- [Background] Kim TH, Kang JW, Kim KH, Kang KW, Shin MS, Jung SY, Kim AR, Jung HJ, Choi JB, Hong KE, Lee SD, Choi SM. Acupuncture for the treatment of dry eye: a multicenter randomised controlled trial with active comparison intervention (artificial teardrops). PLoS One. 2012;7(5):e36638. doi: 10.1371/journal.pone.0036638. Epub 2012 May 17. PMID 22615787
- [Background] Murata A., Uetake A., Ostuka M., Takasawa Y., Proposal of an index to evaluate visual fatigue induced during visual display terminal tasks. International Journal of Human-Computer Interaction 13(3): 305-321, 2001.
- [Background] Wu H.C., Chiu M.C., Jian J.H., Evaluation of Four Eyestrain Recovery Methods for Visual Display Terminal Workers, Communications in Computer and Information Science 617: 536-541, 2016.
- [Background] Nagashima Y., Effect of autonomic nervous activity of the application of heat- and steam- generating sheets to the eyes [in Japanese]. Jpn J Auton Nervous Syst, 43 260-268, 2006.
- [Background] Ochiai R., Moist heat stimulation influence on electroencephalograms and the autonomic nervous system [in Japanese]. Jpn J Auton Nervous Syst, 38: 450-454, 2001.
- [Background] Yang L, Yang Z, Yu H, Song H. Acupuncture therapy is more effective than artificial tears for dry eye syndrome: evidence based on a meta-analysis. Evid Based Complement Alternat Med. 2015;2015:143858. doi: 10.1155/2015/143858. Epub 2015 Apr 16. PMID 25960747